CLINICAL TRIAL: NCT00826683
Title: Detection of Circulating Endothelial Progenitor Cells (EPCs) in Peripheral Blood From Non-small Cell Lung Cancer Patients
Brief Title: Detection of Circulating Endothelial Progenitors Cells (EPCs) in Non-small Cell Lung Cancer (NSCLC)
Acronym: CBNPC:PCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: I08002
Record Dates: First submitted 2009-01-09; First posted 2009-01-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2009-10

CONDITIONS: Non-Small Cell Lung Cancer; Chronic Obstructive Pulmonary Disease
Keywords: Non-small cell lung cancer; Endothelial cell progenitor; Angiogenesis; Vascular endothelial cell growth factor; Healthy control; COPD patients; NSCLC patients
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group of healthy subjects (Other): Control group of healthy subjects : simple blood analysis of EPCs
  Interventions: Biological: Enumeration of endothelial cell progenitor in peripheral blood by flow cytometry, Endothelial cell progenitor characterization by primary cell cultures
- COPD (Active Comparator): COPD: one initial blood sample and simple clinical follow-up
  Interventions: Biological: Enumeration of endothelial cell progenitor in peripheral blood by flow cytometry, Endothelial cell progenitor characterization by primary cell cultures
- NSCLC (Active Comparator): NSCLC: one initial blood sample and usual clinical follow-up
  Interventions: Biological: Enumeration of endothelial cell progenitor in peripheral blood by flow cytometry, Endothelial cell progenitor characterization by primary cell cultures

INTERVENTIONS:
Biological: Enumeration of endothelial cell progenitor in peripheral blood by flow cytometry, Endothelial cell progenitor characterization by primary cell cultures
  Other Names: Characterization of the EPC by the primary cultures,correlation between initial; EPCs and VEGF concentration

SUMMARY:
Bone-marrow-derived progenitor cells (EPCS) play an important role in neovascularization and tumor growth. In lung cancer, angiogenesis is an important event in mechanisms of tumor proliferation and metastasis. Recent evidences suggest that EPCS can be recruited and differentiate in mature endothelial cells to form new blood vessels. The role of EPCs in NSCLC is unclear. In contrast, angiogenic drugs are proposed combined to systemic chemotherapy in NSCLC. The aim of this study is to identify EPCs in peripheral blood from patients with NSCLC, by comparison to Chronic Pulmonary Obstructive Disease (COPD), an inflammatory disease.

DETAILED DESCRIPTION:
The aim of this study is to study blood circulating levels bone-marrow-derived progenitor cells (EPCS).

In a first phase, EPCs will be detected in healthy non-smokers volunteers to validate flow cytometry method (n=25). In addition, EPC will e characterized by primary cultures to analyze EPC-specific markers.

In a second phase, EPCs will detect in peripheral blood from 50 patients with Chronic Obstructive Pulmonary Disease (COPD) and 50 patients with non-small cell lung cancers (NSCLC). Primary cultures will be made to confirm EPCS isolation.

Methods: EPCs will be numerated by flow cytometry using CD133, CD146, CD34, CD45 and VEGFR2 antibodies. Primary cultures will be used to identify EPCs at 5-days culture by the same markers. In addition, for BPCO et NSCLC patients, Vascular endothelial cell growth factor (VEGF) concentration will be measured in peripheral sera by ELISA commercial test.

Overall survival will be analyzed for NSCLC in function of initial EPCs concentration. Correlation will be studied between initial VEGF serum concentration and EPCs level.

This study focus on the possibility that EPC determination in peripheral blood could be used as a surrogate marker of standard or antiangiogenic treatment in NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Signed written consent
* Subject > 18 year old
* No precedent therapy for cancer
* Non-smoker healthy subject or current smoker COPD patients or NSCLC patients

Exclusion Criteria:

* Small-cell lung cancer patient
* Radiotherapy, chemotherapy or target therapy for NSCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Number of EPCs in peripheral blood from NSCLC patients. Comparison with healthy non-smokers patients and smokers with COPD. | at the end of the first step of the study (2 months after the beguening of the study)

SECONDARY OUTCOMES:
Characterization of EPCs by primary cultures. Correlation between initial EPCs and VEGF concentration in COPD and NSCLC patients Overall survival in NSCLC patients in relation to EPCs initial numeration | at he end of the study (10 months after the beguening of the study)

CONTACTS AND LOCATIONS:
Overall Officials: Boris MELLONI, Professor, Principal Investigator — Service de pneumologie,chu Limoges
Locations (1):
- CHU limoges, Limoges, Limoges, France